CLINICAL TRIAL: NCT02198170
Title: A Pharmacokinetic Study to Assess the Influence of Simultaneous CYP3A4 and P-glycoprotein Inhibition on E7080 Pharmacokinetics Following Single Dose Oral Administration of 5 mg E7080 to Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: E7080-A001-004
Record Dates: First submitted 2014-07-21; First posted 2014-07-23 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers
MeSH Terms: interventions — lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ketoconazole-placebo (Experimental): Treatment Period 1: 400 mg ketoconazole orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period Treatment Period 2: Placebo orally once daily + single oral dose of 5 mg lenvatinib of fifth day on 19-day treatment period
  Interventions: Drug: ketoconazole-placebo
- placebo-ketoconazole (Experimental): Treatment Period 1: Placebo orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period Treatment Period 2: 400 mg ketoconazole orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period
  Interventions: Drug: placebo-ketoconazole

INTERVENTIONS:
Drug: ketoconazole-placebo — Treatment Period 1: 400 mg ketoconazole orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period. Treatment Period 2: Placebo orally once daily + single oral dose of 5 mg lenvatinib of fifth day on 19-day treatment period.
  Other Names: E7080
  Arms: ketoconazole-placebo
Drug: placebo-ketoconazole — Treatment Period 1: Placebo orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period Treatment Period 2: 400 mg ketoconazole orally once daily + single oral dose of 5 mg lenvatinib on fifth day of 19-day treatment period
  Other Names: E7080
  Arms: placebo-ketoconazole

SUMMARY:
The purpose of this study is to assess the influence of simultaneous CYP3A4 and p-glycoprotein inhibition on lenvatinib pharmacokinetics following a single oral dose of 5 mg lenvatinib.

DETAILED DESCRIPTION:
This is a single-center, randomized, open-label, two-period, crossover study consisting of two phases: Prerandomization and Randomization. The Prerandomization Phase will have two periods: Screening and Baseline 1. The Randomization Phase will have two periods: Treatment Period 1 and Treatment Period 2 with a Baseline 2 assessment prior to Treatment Period 2. In the Randomization Phase, subjects will be randomized to one of two possible treatment sequences (placebo/ketoconazole or ketoconazole/placebo). Ketoconazole 400 mg or placebo will be orally administered once daily for the first four days of each treatment period. On the fifth day of each treatment period, in addition to ketoconazole/placebo, 5 mg lenvatinib will be orally administered. Ketoconazole/placebo administration will then continue for 13 additional days. Subjects are crossed over from Treatment Period 1 to Treatment Period 2 after a 2-week washout.

ELIGIBILITY:
Inclusion Criteria

1. Non-smoking (i.e., no use of nicotine or nicotine containing products within the past 3 months), male or female subjects, age greater than or equal to 18 years and less than or equal to 55 years
2. Body mass index (BMI) greater than or equal to 18 and less than or equal to 30 kg/m2 at screening
3. All females must have a negative serum and urine B-hCG test result at Screening and Baseline. Females of child-bearing potential must agree to use a medically acceptable method of contraception (e.g., abstinence; a highly effective method such as an intrauterine device [IUD], condom + spermicide or condom + diaphragm with spermicide, a contraceptive implant, an oral contraceptive; or have a vasectomized partner) throughout the entire study period and for 30 days after study drug discontinuation. The only subjects who will be exempt from this requirement are postmenopausal women (defined as greater than age 50 and at least 12 months of amenorrhea) or subjects who have been sterilized surgically or who are otherwise proven sterile (e.g., bilateral tubal ligation with surgery at least 6 months prior to dosing, hysterectomy, or bilateral oophorectomy with surgery at least 2 months prior to dosing). All women who are of reproductive potential and who are using hormonal contraceptives must have been on a stable dose of the same hormonal contraceptive product for at least 12 weeks prior to dosing and must continue to use the same contraceptive during the study and for 30 days after study drug discontinuation.
4. Male subjects who are not abstinent or have undergone a successful vasectomy, who are partners of women of childbearing potential must use, or their partners must use a highly effective method of contraception (e.g., condom + spermicide, condom + diaphragm with spermicide, IUD) starting for at least one menstrual cycle prior to starting study drug(s) and throughout the entire study and for 30 days after the last dose of study drug. Those with partners using hormonal contraceptives must also be using an additional approved method of contraception (as described previously).
5. Provide written informed consent
6. Are willing and able to comply with all aspects of the protocol

Exclusion Criteria

1. Subjects who had a clinically significant illness that required medical treatment within 8 weeks or a clinically significant infection within 4 weeks of dosing
2. Subjects with a disease that may influence the outcome of the study; such as psychiatric disorders and disorders of the gastrointestinal tract, liver, kidney, respiratory system, endocrine system, hematological system, neurological system, or cardiovascular system, or subjects who have a congenital abnormality in metabolism within 4 weeks prior to dosing
3. Subjects with a history of gastrointestinal surgery (hepatectomy, nephrotomy, digestive organ resection, etc.) that may affect pharmacokinetic profiles of lenvatinib
4. Subjects with a known history of clinically significant drug or food allergies or presently experiencing significant seasonal allergy
5. Subjects who experienced a weight loss or gain of greater than 10% between screening and prior to dosing
6. Subjects with any clinically abnormal symptom or organ impairment found on medical history, symptoms/signs, vital signs, ECG finding, or laboratory test results which require medical treatment
7. Subjects with a QTc interval greater than 450 ms at screening or check-in
8. Subjects with hemoglobin level less than 12.0 g/dL
9. Subjects who had a positive result from human immunodeficiency virus (HIV) or hepatitis C virus antibody (HCVAb) screening tests, or clinical evidence of active viral Hepatitis A or B
10. Subjects with a known or suspected history of drug or alcohol misuse within 6 months prior to screening, or a positive urine drug or alcohol test at screening or baseline
11. Subjects who have consumed caffeinated beverages within 72 hours prior to baseline
12. Subjects who have taken dietary supplements, juice, or herbal preparations or other foods or beverages that may affect various drug metabolizing enzymes and transporters [e.g., alcohol, grapefruit, grapefruit juice, grapefruit-containing beverages, apple or orange juice), vegetables from the mustard green family (e.g., kale, broccoli, watercress, collard greens, kohlrabi, brussel sprouts, mustard), and charbroiled meats] within 2 weeks prior to dosing
13. Subjects who have taken herbal preparations containing St. John's Wort within 4 weeks prior to dosing
14. Subjects who have taken prescription drugs within 4 weeks prior to screening (however, use of prescription contraceptive products is permitted)
15. Subjects who have taken over-the-counter (OTC) medications within 2 weeks prior to dosing
16. Subjects who have participated in another clinical trial of an investigational drug or device within 4 weeks prior to dosing
17. Subjects who have received blood products within 4 weeks, or donated blood within 8 weeks, or donated plasma within 1 week of dosing
18. Subjects who have engaged in heavy exercise within 2 weeks prior to check-in (e.g., marathon runners, weight lifters, etc.)
19. Subjects who are unwilling or unable to abide by the requirements of the study
20. Subjects who have any condition that would make him/her, in the opinion of the investigator, unsuitable for the study or who, in the opinion of the investigator, are not likely to complete the study for any reason
21. Known intolerance to the study drugs or any of the excipients
22. Females who are either pregnant or lactating

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2011-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of CYP3A4 and p-glycoprotein inhibition on lenvatinib: Cmax | Baseline 1 (Day -1) and 2 (Day 33); Treatment period 1 and 2: Predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, 120, 144, 168, 240, 288, and 336 hours post dose
Pharmacokinetics of CYP3A4 and p-glycoprotein inhibition on lenvatinib: AUC(0-t) | Baseline 1 (Day -1) and 2 (Day 33); Treatment period 1 and 2: Predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, 120, 144, 168, 240, 288, and 336 hours post dose
Pharmacokinetics of CYP3A4 and p-glycoprotein inhibition on lenvatinib: AUC(0-inf) | Baseline 1 (Day -1) and 2 (Day 33); Treatment period 1 and 2: Predose and at 0.5, 1, 2, 3, 4, 8, 12, 16, 24, 48, 72, 96, 120, 144, 168, 240, 288, and 336 hours post dose

SECONDARY OUTCOMES:
Safety as Measured by Outcome of Adverse Events | Screening, Up to Day 52
Safety as Measured by Laboratory Values | Screening, Up to Day 52
Safety as Measured by Vital Signs | Screening, Up to Day 52
Safety as Measured by ECGs | Screening, Up to Day 52
Safety as Measured by Physical Examination | Screening, Up to Day 52

CONTACTS AND LOCATIONS:
Locations (1):
- Tacoma, Washington, United States